CLINICAL TRIAL: NCT06732349
Title: Urinary Tubular Biomarkers for Chronic Kidney Disease
Acronym: U-Tube 1
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Full Professor of Nephrology, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2024-0505 - U-Tube 1
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Stage 3
Keywords: biomarker; disease progression; chronic kidney disease; tubular function and injury; urine; risk assessment; personalized medicine
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spot urine samples which are collected for routine clinical evaluation at the outpatient department
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Urinary tubular test panel — The urinary tubular test panel will be applied to urine samples that are collected as part of the routine outpatient follow-up. Its predictive power for CKD progression will be assessed. The results of the tubular test panel will not influence the treatment of the patients. They will remain under standard outpatient treatment throughout the study.

SUMMARY:
Currently used tests for chronic kidney injury only assess the function of one part of the kidney: the filter called the glomerulus. The other part, called the tubule, is disregarded. Based on many previous studies, the investigators have good reason to assume that a better prediction of the course of chronic kidney disease by testing tubular function will be possible. This is important, for example, when patients need to be treated with kidney-protecting drugs.

DETAILED DESCRIPTION:
Rationale Chronic kidney disease (CKD) is a common and progressive condition that affects over 800 million people worldwide and is now one of the leading causes of mortality. The kidney consists of filters and tubules, but diagnosis of progressive CKD is currently based on filter function alone (estimated glomerular filtration rate (eGFR) and albuminuria). However, it is tubular injury that drives CKD progression, and it is the tubule that is targeted by recently developed kidney-protective treatments. We hypothesize that a high-throughput tubular test panel, consisting of urine supersaturation and urinary extracellular vesicle (uEV) biomarkers, improves the prediction of CKD progression thereby enabling the early initiation of kidney-protective treatment.

Objective(s) To develop a high-throughput tubular test panel, consisting of urine supersaturation and uEV biomarkers, that improves the prediction of CKD progression.

Study type Prospective diagnostic trial.

Study population Adult patients with CKD stage G3 (eGFR 30-59 ml/min/1.73 m2).

Methods Urine samples are already collected as part of the standard of care and will be divided for measurement of albuminuria (standard of care) and urine supersaturation and uEV biomarkers (this project). The performance of the tubular test panel will be analyzed by comparing it to that of the existing Kidney Failure Risk Equation.

Burden and risks The diagnostic tests will be performed on a urine sample that is already collected as part of routine clinical care. Therefore, these diagnostic procedures do not pose an additional risk or burden.

Recruitment and consent Participants will be recruited from the Department of Internal Medicine outpatient clinics. For all study participants written informed consent will be obtained. The informed consent will include the approval (yes/no) to store samples for secondary use.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 3 (eGFR 30-59ml/min)

Exclusion Criteria:

* Active glomerulonephritis treated with immunosuppression
* Kidney transplant recipient
* Current treatment with chemo- or immunotherapy for malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≤18 years) with CKD stage 3, treated at the Internal Medicine outpatient department of the Erasmus MC university hospital (convenience sampling).
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
CKD Progression | 3 years
  Rate of participants that reach the composite of 30% reduction in estimated glomerular filtration rate (CKD-EPI creatinine-based) and/or the initiation of kidney replacement therapy (dialysis or kidney transplantation)

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR, Analytic Code